CLINICAL TRIAL: NCT07206914
Title: Geographic Analysis of Cancer Patients' Residences at Delafontaine Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0116_ONCOLOGIE
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms; Oncology Service; Health Services Accessibility; Health Inequalities; Residence Characteristics; Transportation of Patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study looks at where cancer patients treated at Delafontaine Hospital live and how far they have to travel for care. By mapping patients' home addresses (anonymized), the research will show how distance, transportation, and social factors affect access to cancer treatments and support services. The goal is to better understand inequalities in access to care and to improve patient support in the future.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients treated for cancer in the oncology department of Delafontaine Hospital since January 1, 2020.

Exclusion Criteria:

- Patients whose cancer treatment in the oncology department was completed before 2020.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be selected from the population of patients treated for cancer in the oncology department of Delafontaine Hospital, located in Seine-Saint-Denis (93), France. This population includes adult patients receiving chemotherapy, radiotherapy, targeted therapies, immunotherapy, or supportive care as part of their cancer management. Since Delafontaine Hospital is a public hospital in a densely populated and socioeconomically diverse area of the Paris region, the patient population is expected to reflect a wide range of social, cultural, and economic backgrounds, including a high proportion of individuals from immigrant communities. This diversity provides a valuable context for studying inequalities in geographic accessibility to oncology care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Median travel time (minutes) from the patient's place of residence (IRIS centroid) to Delafontaine Hospital by the patient's usual mode of transport for oncology appointments. | Assessed up to 5 years after first inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France, France